CLINICAL TRIAL: NCT07353957
Title: A Phase 2 Study to Investigate the Safety and Efficacy of Petosemtamab in Adults With Metastatic Non-Small Cell Lung Cancer in Combination With Pembrolizumab as First-Line Treatment
Brief Title: Study to Investigate Petosemtamab in Adults With Metastatic Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merus B.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCLA-158-CL04
Record Dates: First submitted 2026-01-16; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer - Non Small Cell Squamous; Lung Cancer - Non Small Cell Non-Squamous
Keywords: squamous; lung cancer; non-squamous lung cancer; petosemtamab
MeSH Terms: conditions — Lung Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- First line squamous non-small cell lung cancer patients (Experimental)
  Interventions: Combination Product: Petosemtamab + Pembrolizumab
- First line non-squamous non-small cell lung cancer patients (Experimental)
  Interventions: Combination Product: Petosemtamab + Pembrolizumab

INTERVENTIONS:
Combination Product: Petosemtamab + Pembrolizumab — Petosemtamab + Pembrolizumab

SUMMARY:
The study will test the efficacy and safety of petosemtamab in combination with Pembrolizumab in first line patients with squamous non-small cell lung cancer and non-squamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent and is willing and able to comply with all study procedures and contraception requirements
* Age ≥ 18 years at the signing of ICF
* At least 1 measurable lesion as defined by RECIST 1.1
* ECOG performance status of 0 or 1
* Life expectancy ≥ 12 weeks, in the opinion of the Investigator
* Adequate hematologic function
* Creatinine clearance ≥ 60 mL/min calculated according to the Cockroft and Gault formula
* Adequate liver function
* Serum albumin ≥ 3 g/dL
* Serum magnesium and corrected calcium, Grade ≤ 1 alteration
* Participants of childbearing potential must agree to use highly effective contraception methods for the duration of study participation
* Histologically confirmed metastatic (Stage IV) sqNSCLC with PD-L1 TPS ≥ 50%
* No prior systemic treatment for metastatic disease
* Testing is required per local SOC and availability of testing to document absence of actionable genomic tumor aberrations
* Histologically confirmed metastatic (Stage IV) non-squamous NSCLC with PD-L1 TPS ≥ 50%

Exclusion Criteria:

* Has untreated CNS metastases and/or carcinomatous meningitis
* Participation in an interventional clinical study with any investigational drug within 4 weeks prior to the first dose of study treatment OR participation in any clinical study with petosemtamab at any time prior to the first dose of study treatment, regardless of whether petosemtamab was received
* Participants who received prior treatment with a PD-(L)1 inhibitor
* Participants who have received prior systemic chemotherapy, targeted or biological antineoplastic therapy for metastatic NSCLC
* Any systemic anticancer therapy within 4 weeks prior to the first dose of study treatment
* Major surgery or radiotherapy within 3 weeks prior to the first dose of study treatment. Participants who received prior radiotherapy to ≥ 25% of bone marrow are not eligible, regardless of when it was received.
* Persistent Grade > 1 clinically significant toxicities related to prior antineoplastic therapies using NCI-CTCAE v5.0
* History of hypersensitivity reaction to any of the excipients of petosemtamab or pembrolizumab
* Unstable angina; history of congestive heart failure of Class II-IV New York Heart Association criteria or serious cardiac arrhythmia requiring treatment (except atrial fibrillation, paroxysmal supraventricular tachycardia); or history of myocardial infarction within 6 months prior to the first dose of study treatment
* History of prior malignancies within the last 5 years, with the exception of excised local cancer
* Current dyspnea at rest of any origin or other diseases requiring continuous oxygen therapy, including participants with a history of ILD (eg, pneumonitis or pulmonary fibrosis) or evidence of ILD on baseline chest CT scan
* Current serious illness or medical condition, including but not limited to uncontrolled active infection and clinically significant pulmonary, metabolic, or psychiatric disorders
* Known infectious disease
* Participants who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2031-02-27 (Estimated)

PRIMARY OUTCOMES:
Objective response rate per investigator assessment | Up to 4.5 years
  ORR was defined as the proportion of participants who had a complete response (CR) or partial response (PR) per RECIST v1.1.

SECONDARY OUTCOMES:
Duration of response per Investigator assessment | Up to 4.5 years
  For participants with a confirmed CR or PR per RECIST v1.1, DOR was defined as the time from the date of first documented response of CR or PR per RECIST v1.1 to the date of first documented progression or death due to underlying cancer.
Disease control rate as per investigator assessment | Up to 4.5 years
  DCR is defined as the proportion of participants with CR or PR or stable disease (SD) per RECIST 1.1.
Clinical Benefit Rate as per investigator assessment | Up to 4.5 years
  CBR was defined as the proportion of participants with a CR or PR, or SD lasting ≥24 weeks per RECIST v1.1
Progression free survival as per investigator assessment | Up to 4.5 years
  PFS was defined as the time from first dose to the first documented disease progression per RECIST v1.1 or death due to any cause.
Overall survival | Up to 4.5 years
  OS was defined as the time from first dose to death due to any cause.
Number of participants who experienced on treatment adverse events | Up to 4.5 years
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. Severity of AEs will be graded according to the NCI CTCAE version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening and Grade 5: death related to adverse event.
Concentrations of petosemtamab predose and at end of infusion | Up to 6-12 months
  Predose and end of infusion plasma concentrations as measured from all individual plasma concentrations.
Incidence and serum titers of anti-drug antibodies (ADAs) against petosemtamab | Up to 6-12 months
  The frequency and proportion of participants developing anti-drug antibodies.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Tennessee Site 2, Chattanooga, Tennessee
  - Tennessee Site 1, Nashville, Tennessee
  - Virginia Site 1, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No